CLINICAL TRIAL: NCT05527821
Title: An Exploratory Clinical Study of Short Course Radiotherapy Combined With Surufatinib and Sintilimab in the Treatment of Relapsed and Refractory Advanced Solid Tumors
Brief Title: Study of Surufatinib Combined With Sintilimab and SCRT in Advanced Solid Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaorong Dong, Director, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-ST101
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Unresectable Advanced Solid Tumors; Biliary Tract Tumors, Gastric Cancer, Small Cell Lung Cancer
MeSH Terms: conditions — Stomach Neoplasms; Small Cell Lung Carcinoma | interventions — surufatinib; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surufatinib Combined With Sintilimab and SCRT (Experimental)
  Interventions: Drug: Surufatinib; Drug: Sintilimab; Radiation: Short course radiotherapy

INTERVENTIONS:
Drug: Surufatinib — Surufatinib 250mg will be taken orally once daily continuously on a 21-day cycle
Drug: Sintilimab — Sintilimab 200mg will be intravenously administered on Day 1 of each cycle
Radiation: Short course radiotherapy — 5Gy*5F short course radiotherapy will be delivered

SUMMARY:
An exploratory clinical study of short course radiotherapy combined with surufatinib and sintilimab in the treatment of relapsed and refractory advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years (including 18 and 75 years), both genders;
2. Unresectable malignant tumors confirmed by histology or cytology (mainly biliary tract tumors, gastric cancer, small cell lung cancer, and other tumor types were included as appropriate), which failed at least after first-line standard treatment;
3. The lesions can be clearly evaluated by imaging;
4. Expected survival ≥ 12 weeks;
5. No serious abnormalities of blood system, heart, lung, liver, kidney function or immune deficiency;
6. Laboratory tests (without blood transfusion within 14 days) shall meet the following requirements:
7. If a fertile man or woman is willing to use contraception during the trial;
8. Physical status score ECOG 0-1;
9. Patients or their family members agreed to participate in the study and signed the informed consent form;

Exclusion Criteria:

1. Previous treatment with anti-VEGF/VEGFR-targeted drugs, such as surufatinib; Or previous treatment with anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs or another stimulatory or synergistic inhibition of T-cell receptors (including but not limited to CTLA-4, OX-40, LAG-3, CD137, etc.);
2. Women who are breast feeding, pregnant or preparing to become pregnant;
3. Corticosteroids (dose equivalent to prednisone & GT; 10 mg/ day) or other immunosuppressive therapy;
4. Active, known or suspected autoimmune diseases or before 2 years of the history of the disease (in nearly 2 years can be treated as system of vitiligo, psoriasis, hair loss, or graves disease, need only thyroid hormone replacement therapy for hypothyroidism and only need insulin replacement therapy in patients with type 1 diabetes can group);
5. Allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation; Persons with HIV infection or active hepatitis b or c (active hepatitis b reference: HBV DNA≥1×104 copies /ml or ≥2000IU/ml; Active hepatitis C reference: HCV RNA≥1×103 copies /ml);
6. Interstitial lung disease (including past history and current condition), such as interstitial pneumonia, pulmonary fibrosis, or evidence of ILD on baseline chest CT or MRI;
7. Allergic constitution and multiple drug allergy;
8. Patients judged by other investigators to be unable to tolerate chemotherapy or not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | From Baseline to primary completion date, about 24 months
  A duration from the date of initial treatment to disease progression or death of any cause

SECONDARY OUTCOMES:
Objective response rate (ORR) | From Baseline to primary completion date, about 24 months
  The incidence of confirmed complete response or partial response
Disease Control Rate | From Baseline to primary completion date, about 24 months
  The incidence of complete response, partial response and stable disease
Overall survival (OS) | From the time of enrollment to death caused by any reason
  From Baseline to primary completion date, about 24 months
The incidence of adverse events | From Baseline to primary completion date, about 24 months
  The safety and tolerability of Surufatinib will be evaluated based on adverse events data

CONTACTS AND LOCATIONS:
Locations (1):
- Union hospital, Wuhan, Hubei, China